CLINICAL TRIAL: NCT01440595
Title: A Randomized, Partially Double-Blind, Active-Controlled, Dose-Ranging Estimation Study to Evaluate the Safety, Tolerability, and Efficacy of Different Regimens of MK-5172 When Administered Concomitantly With Pegylated-Interferon and Ribavirin in Treatment-Naive Patients With Chronic Genotype 2 or 3 Hepatitis C Virus Infection
Brief Title: Grazoprevir (MK-5172) With Peg-Interferon and Ribavirin in Participants With Chronic Genotype 2 or 3 Hepatitis C (MK-5172-012)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Preliminary results of MK-5172 PN003 (NCT01353911) suggested a possible dose relationship to elevated transaminase levels in treatment with grazoprevir.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5172-012; 2011-003299-36 (EudraCT Number)
Record Dates: First submitted 2011-09-22; First posted 2011-09-26 (Estimated); Results first posted 2016-03-04 (Estimated); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — grazoprevir; peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Grazoprevir 200 mg + Peg-IFN + RBV (Experimental): Grazoprevir 200 mg in combination with Peg-IFN and RBV for 12 weeks.
  Interventions: Drug: Grazoprevir; Drug: Peginterferon alfa-2b (Peg-IFN); Drug: Ribavirin (RBV)
- Grazoprevir 400 mg + Peg-IFN + RBV (Experimental): Grazoprevir 400 mg in combination with Peg-IFN and RBV for 12 weeks.
  Interventions: Drug: Grazoprevir; Drug: Peginterferon alfa-2b (Peg-IFN); Drug: Ribavirin (RBV)
- Placebo + Peg-IFN + RBV (Placebo Comparator): Placebo to grazoprevir in combination with Peg-IFN and RBV for 12 weeks, followed by open-label Peg-IFN and RBV for an additional 12 weeks.
  Interventions: Drug: Placebo to Grazoprevir; Drug: Peginterferon alfa-2b (Peg-IFN); Drug: Ribavirin (RBV)
- Grazoprevir 800 mg + Peg-IFN + RBV (Experimental): Grazoprevir 800 mg in combination with Peg-IFN and RBV for 12 weeks.
  Interventions: Drug: Grazoprevir; Drug: Peginterferon alfa-2b (Peg-IFN); Drug: Ribavirin (RBV)

INTERVENTIONS:
Drug: Grazoprevir — Grazoprevir 100 mg tablets once daily for 12 weeks.
  Other Names: MK-5172
  Arms: Grazoprevir 200 mg + Peg-IFN + RBV; Grazoprevir 400 mg + Peg-IFN + RBV; Grazoprevir 800 mg + Peg-IFN + RBV
Drug: Placebo to Grazoprevir — Placebo to Grazoprevir once daily for 12 weeks
  Arms: Placebo + Peg-IFN + RBV
Drug: Peginterferon alfa-2b (Peg-IFN) — Peg-IFN weekly subcutaneous injection at 1.5 mcg/kg/week for 12 or 24 weeks
  Other Names: PegIntron®, SCH 054031
Drug: Ribavirin (RBV) — Ribavirin 200 mg capsules twice daily at a dose of 600 mg to 1400 mg based on weight for 12 or 24 weeks
  Other Names: Rebetol®, SCH 018908

SUMMARY:
This study will evaluate the safety, tolerability, and antiviral activity of grazoprevir (MK-5172) when administered concomitantly with peg-interferon alfa-2b (Peg-IFN) and ribavirin (RBV) to treatment-naïve participants with chronic genotype 2 (GT2) or genotype 3 (GT3) hepatitis C virus (HCV) infections.

ELIGIBILITY:
Inclusion Criteria:

* Body weight ≥ 88 lbs and ≤ 275 lbs
* Documented chronic Hepatitis C (CHC) GT2 or GT3 infection
* No known cirrhosis
* Agrees to use two acceptable methods of birth control during study and through 6 months after last dose of study drug
* Chest X-ray within the last 6 months
* Eye exam within the last 6 months

Exclusion Criteria:

* Known to be human immunodeficiency virus (HIV) positive or co-infected with active hepatitis B virus (positive for Hepatitis B surface antigen)
* Prior approved or investigational treatment for hepatitis C
* Evidence of hepatocellular carcinoma
* Diabetic and/or high blood pressure with clinically significant eye exam findings
* Pre-existing psychiatric condition
* Clinical diagnosis of abuse of certain substances within specified timeframes
* Known medical condition that could interfere with participation
* Active or suspected cancer within the last 5 years
* Female who is pregnant, breastfeeding, or expecting to conceive or donate eggs
* Male who is planning to impregnate partner or donate sperm
* Male with a pregnant female partner
* Chronic hepatitis not caused by HCV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-11-28 (Actual); Primary Completion 2012-05-01 (Actual); Study Completion 2012-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=5172-012&kw=5172-012&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were randomized to the Grazoprevir 800 mg + Peg-IFN + RBV arm.
Groups:
- Grazoprevir 200 mg + Peg-IFN + RBV: Grazoprevir 200 mg once daily by mouth in combination with Peg-IFN and RBV for 12 weeks.
- Grazoprevir 400 mg + Peg-IFN + RBV: Grazoprevir 400 mg once daily by mouth in combination with Peg-IFN and RBV for 12 weeks.
- Placebo + Peg-IFN + RBV: Placebo to grazoprevir once daily by mouth in combination with Peg-IFN and RBV for 12 weeks, followed by open-label Peg-IFN and RBV for an additional 12 weeks.
Period: Overall Study
Arm/Group | Grazoprevir 200 mg + Peg-IFN + RBV | Grazoprevir 400 mg + Peg-IFN + RBV | Placebo + Peg-IFN + RBV
Started | 1 | 3 | 1
Completed | 0 | 0 | 0
Not Completed | 1 | 3 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Study terminated by sponsor. | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Five participants were randomized as indicated in the Participant Flow Module, but only 3 participants were treated. Baseline Characteristics are presented only for treated participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Grazoprevir 400 mg + Peg-IFN + RBV | Placebo + Peg-IFN + RBV | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (7.8) | 51.0 (0.0) | 44.0 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Complete Early Virologic Response (cEVR) in the Grazoprevir Treatment Arms
Description: cEVR was defined as undetectable hepatitis C virus (HCV) ribonucleic acid (RNA) at Week 12. HCV RNA was measured using the Roche COBAS® Taqman® HCV Test, v.2.0 assay.
Time Frame: Week 12
Population: The Full Analysis Set (FAS) population includes all randomized participants who received at least 1 dose of study treatment. No participants completed treatment, and no analyses were conducted for this study due to early termination.
Arm/Group | Grazoprevir 400 mg + Peg-IFN + RBV | Placebo + Peg-IFN + RBV
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Time to First Achievement of Undetectable HCV Ribonucleic Acid (RNA)
Description: Time to first achievement of undetectable HCV RNA was determined by measuring HCV RNA at Treatment Days 1, 3, and 7; Treatment Weeks 2, 4, 8, 12, 16, 20, and 24; as well as Follow-up Weeks 4, 12, and 24. HCV RNA was measured using the Roche COBAS® Taqman® HCV Test, v2.0 assay.
Time Frame: Baseline to Week 12 for Grazoprevir treatment arms, Week 24 for Placebo arm
Population: as for outcome 1
Arm/Group | Grazoprevir 400 mg + Peg-IFN + RBV | Placebo + Peg-IFN + RBV
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants Achieving Rapid Viral Response (RVR)
Description: RVR was defined as undetectable HCV RNA at Week 4. HCV RNA was measured using the Roche COBAS® Taqman® HCV Test, v2.0 assay.
Time Frame: Week 4
Population: as for outcome 1
Arm/Group | Grazoprevir 400 mg + Peg-IFN + RBV | Placebo + Peg-IFN + RBV
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Participants Achieving Sustained Viral Response 12 Weeks After Completion of Therapy (SVR12)
Description: SVR12 was defined as undetectable HCV RNA 12 weeks after completion of study therapy. HCV RNA was measured using the Roche COBAS® Taqman® HCV Test, v2.0 assay.
Time Frame: Week 24 for Grazoprevir treatment arms, Week 36 for Placebo arm
Population: as for outcome 1
Arm/Group | Grazoprevir 400 mg + Peg-IFN + RBV | Placebo + Peg-IFN + RBV
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants Achieving Sustained Viral Response 24 Weeks After Completion of Therapy (SVR24)
Description: SVR24 was defined as undetectable HCV RNA 24 weeks after completion of study therapy. HCV RNA was measured using the Roche COBAS® Taqman® HCV Test, v2.0 assay.
Time Frame: Week 36 for Grazoprevir treatment arms, Week 48 for Placebo arm
Population: as for outcome 1
Arm/Group | Grazoprevir 400 mg + Peg-IFN + RBV | Placebo + Peg-IFN + RBV
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Participants Achieving Undetectable HCV RNA at Week 12 in the Placebo Arm
Description: HCV RNA was measured using the Roche COBAS® Taqman® HCV Test, v2.0 assay.
Time Frame: Week 12
Population: as for outcome 1
Arm/Group | Grazoprevir 400 mg + Peg-IFN + RBV | Placebo + Peg-IFN + RBV
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants Achieving Complete Early Virologic Response (cEVR) at Week 24 in the Placebo Arm
Description: cEVR was defined as undetectable hepatitis C virus (HCV) ribonucleic acid (RNA) at Week 24 (i.e., after 12 weeks of placebo + 12 weeks of grazoprevir treatment). HCV RNA was measured using the Roche COBAS® Taqman® HCV Test, v2.0 assay.
Time Frame: Week 24
Population: as for outcome 1
Arm/Group | Grazoprevir 400 mg + Peg-IFN + RBV | Placebo + Peg-IFN + RBV
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Non-serious AEs were collected up to Week 26 and serious AEs (SAEs) were collected up to Week 48.
Arm/Group | Grazoprevir 400 mg + Peg-IFN + RBV | Placebo + Peg-IFN + RBV
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Grazoprevir 400 mg + Peg-IFN + RBV (N=2) | Placebo + Peg-IFN + RBV (N=1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 1 (1)
Irritabilty (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Skeletal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Restless leg syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation.